CLINICAL TRIAL: NCT07163364
Title: A Single-arm Phase III Clinical Study to Evaluate the Efficacy and Safety of Hydroxocobalamin Chloride Injection in Participants With Methylmalonic Acidemia (MMA) With Elevated Homocysteine (Cobalamin C Deficiency)
Brief Title: A Study to Evaluate the Effects and Safety of Hydroxocobalamin in Participants With Combined Methylmalonic Academia (cblC Type)
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYH9097-001
Record Dates: First submitted 2025-08-19; First posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-08

CONDITIONS: Methylmalonic Acidemia (MMA)
MeSH Terms: conditions — Methylmalonic acidemia

STUDY DESIGN:
Intervention Model Description: This study is a Single-Center, Single-Arm, open-label, Phase III clinical study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hydroxocobalamin Chloride Injection (Experimental): Hydroxocobalamin Chloride Injection
  Interventions: Drug: Hydroxocobalamin Chloride Injection

INTERVENTIONS:
Drug: Hydroxocobalamin Chloride Injection — 1 - 20 mg per dose, 1 - 5 times per week

SUMMARY:
This study is a Single-Center, Single-Arm, open-label, Phase III clinical study to evaluate the efficacy, safety characteristics of Hydroxocobalamin Chloride Injection (20 mg/mL) for Maintenance Therapy in participants with Methylmalonic Acidemia (MMA) with Elevated Homocysteine (Cobalamin C Deficiency).

ELIGIBILITY:
Inclusion Criteria:

1. Age 6 months (inclusive) to < 18 years at the time of first investigational product administration; both sexes eligible.
2. Confirmed diagnosis of cobalamin C (cbl C)-type methylmalonic acidemia (MMA) fulfilling ALL of the following:

   1. Documented vitamin B12 responsiveness: ≥ 50 % reduction from pre-treatment baseline in plasma C3/C2 ratio and urinary methylmalonic acid following vitamin B12 therapy.
   2. Presence of pathogenic MMACHC gene variants in a participant with MMA associated with hyperhomocysteinemia.
3. Investigator-assessed clinical stability, defined as:

   * No emergency room visits or hospitalizations within 6 months prior to screening for metabolic crises (e.g., electrolyte disturbances, metabolic acidosis, dysglycaemia, multi-organ failure); AND
   * Plasma methylmalonic acid within the normal reference range at screening.
4. Continuous treatment with injectable hydroxocobalamin for ≥ 3 months immediately preceding first dose of study drug.
5. Written informed consent obtained from participant and/or legally authorised representative; willingness and ability to comply with all study visits and procedures.
6. Female participants of childbearing potential (post-menarche) must have a negative serum β-hCG test at screening. All participants of reproductive potential (post-menarche females or males with documented spermarche) must use a highly effective contraceptive method throughout the study and for an appropriate post-study period as defined by local regulations.

Exclusion Criteria:

1. Use of any vitamin B12 preparation other than injectable hydroxocobalamin within 3 months prior to screening.
2. Participation in another clinical trial within 28 days or 5 half-lives of the investigational agent (whichever is longer) before screening initiation, except for screening-only participants who did not receive study drug.
3. Prior liver or kidney transplantation, or any prior cell-based therapy.
4. Any of the following laboratory abnormalities:

   * Hemoglobin < 90 g/L; or
   * Platelet count < 100 × 10⁹/L; or
   * Estimated glomerular filtration rate (eGFR) < 60 mL/min/1.73 m²; or
   * Requirement for dialysis due to renal disease.
5. Evidence of clinically significant hepatic dysfunction defined as:

   1. Alanine aminotransferase (ALT) > 2.0 × upper limit of normal (ULN);
   2. Aspartate aminotransferase (AST) > 2.0 × ULN or total bilirubin > 1.5 × ULN;
   3. Prothrombin time > 1.5 × ULN.
6. Hyperammonemia characterised by blood ammonia ≥ 3 × ULN, or any acute metabolic decompensation (e.g., lethargy, restlessness, somnolence, feeding refusal, or vomiting).
7. Evidence on prior imaging of a space-occupying lesion suspicious for malignancy, or any known history of malignancy.
8. New York Heart Association (NYHA) Class III or IV heart failure, or moderate-to-severe pulmonary hypertension.
9. Clinically significant urolithiasis identified on imaging performed during screening.
10. Presence of any of the following underlying conditions: immunodeficiency, severe malnutrition, congenital heart disease, congenital malformations of the respiratory system, or any clinically significant cardiac, hepatic, pulmonary, or renal disorder; diabetes mellitus; severe hematological disease; uncontrolled epilepsy or other significant central nervous system disorders.
11. History of severe hypersensitivity or known hypersensitivity/intolerance to hydroxocobalamin, structurally related compounds, or any excipients in the investigational product.
12. Any other condition or circumstance that, in the judgment of the investigator, would compromise participant safety, compliance, or data integrity.

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-08-31 (Estimated); Primary Completion 2026-10-08 (Estimated); Study Completion 2027-04-28 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants achieving normalization of plasma or urinary methylmalonic acid levels post-dose. | Week4、Week6、Week10、Week16、Week24

SECONDARY OUTCOMES:
Change from baseline in plasma total homocysteine level. | Day3、Week2、Week4、Week6、Week10、Week16、Week24、Week32、Week40、Week48
Change from baseline in plasma propionylcarnitine (C3), plasma C3/acetylcarnitine (C2) ratio, and urinary methylcitrate. | Day3、Week2、Week4、Week6、Week10、Week16、Week24、Week32、Week40、Week48
Change from baseline in plasma methylmalonic acid concentration. | Day3、Week2、Week4、Week6、Week10、Week16、Week24、Week32、Week40、Week48
Change from baseline in urinary methylmalonic acid excretion. | Day3、Week2、Week4、Week6、Week10、Week16、Week24、Week32、Week40、Week48
Proportion of participants achieving plasma methylmalonic acid levels within the normal reference range. | Week32、Week40、Week48
Proportion of participants achieving urinary methylmalonic acid levels within the normal reference range. | Week32、Week40、Week48
Change from baseline in growth parameters (height). | Week24、Week48
Change from baseline in growth parameters (weight) | Week24、Week48
Change from baseline in growth parameters (head circumference). | Week24、Week48
Change from baseline in Gesell Developmental Scales. | Week24、Week48
  Higher scores means a better outcome.
Change from baseline in Wechsler Intelligence Scale | Week24、Week48
  Higher scores means a better outcome.